CLINICAL TRIAL: NCT03522909
Title: The Center for Peripartum Optimization: An Innovative Approach to Care Coordination
Brief Title: The Center for Peripartum Optimization
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00163559
Record Dates: First submitted 2018-05-01; First posted 2018-05-11 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2020-07

CONDITIONS: High Risk Pregnancy; Multidisciplinary Communication; Communication; Obstetric Complication
Keywords: obstetric anesthesia; telemedicine
MeSH Terms: conditions — Communication | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: We will be reviewing records of parturients seen at Johns Hopkins Hospital in the Center for Peripartum Optimization (CPO) clinic between January 2017 to January 2018
  Interventions: Other: Seen in clinic
- Control: A matched controlled group patients not seen at the CPO clinic

INTERVENTIONS:
Other: Seen in clinic — We will be doing a retrospective chart review of patients seen in the Center for Peripartum Optimization to look for:
  1. Primary outcome variable.
     - Hospital length of stay
  2. Secondary outcome variables.
     * Number of admissions from outside hospitals
     * Adverse outcomes
     * Intensive Care Unit admissions
     * Opioid use
     * NICU admissions
     * Patient satisfaction
     * Cost of inpatient admission
     * Cost of outpatient care
     * Hospital readmissions rate
  Groups: Study

SUMMARY:
In January 2017 investigators started a Center for Peripartum Optimization (CPO) with the aim of optimizing a patient's clinical status in an outpatient setting to minimize unnecessary laboratory tests and studies, costly inpatient consultations, the likelihood of post-surgical adverse events, escalations in level of care, inpatient admissions and readmissions. This research project seeks to evaluate the impact of this innovative concept on patient outcomes during the last 12 months. Investigators will accomplish this by collecting retrospective data from patients' electronic medical records in the intervention group and comparing it to data gathered from a controlled group of patients with similar comorbidities but who were not evaluated at the CPO clinic.

ELIGIBILITY:
Inclusion Criteria:

* Records of all female, obstetric patients of child-bearing age who were evaluated in the Center for Peripartum Optimization during the period between January 2017 and January 2018.
* Controlled group will include parturients with match high risk comorbidities or history of nonobstetric surgery during pregnancy who delivered at Johns Hopkins Hospital (JHH) during July 1, 2016 - Dec 31, 2016
* Patients with any one or more of these high risk comorbidities:
* Complex spine pathologies (Scoliosis, vertebral fusion, disc disease, spinal canal defects, neuropathies, and nerve disease, etc.)
* Neurological pathology (Cerebral ischemia, tumor, increased intracranial pressure, cerebral vascular disease, etc.)
* Cardiac disease (Congenital, valvular, pulmonary hypertension, cardiomyopathy, ischemic disease, arrhythmia, etc.)
* Pulmonary disease (History of pulmonary embolism, interstitial lung disease, severe asthma, cancer, etc.)
* Morbid Obesity (Obstructive Sleep Apnea, equipment considerations)
* Hematologic Disorders (Thrombophilias, coagulopathies, patients on anticoagulation)
* Cancer
* Abnormal placentation (Previa, accreta / increta / percreta)
* Anesthetic concerns (Airway abnormalities, history of adverse anesthetic reactions or experiences (i.e. recall, anaphylaxis))
* Fetal therapy patients requiring specialized management (Ex utero intrapartum treatment (EXIT), Fetoscopic endotracheal occlusion (FETO), Twin-to-twin transfusion syndrome (TTTS), Percutaneous Umbilical Blood Sampling (PUBS), etc.)
* Chronic Pain

Exclusion Criteria:

* Records of CPO participating parturients outside the specified timeframe.
* Records of obstetric patients of child-bearing age without high-risk comorbid conditions described in inclusion criteria.
* Records of patients seen in CPO clinic that did not deliver at our institution

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Pregnant patients
Study Population: This will be a retrospective study design utilizing the Johns Hopkins Hospital (JHH) electronic medical record system (EMR) "EPIC". We will be reviewing records of parturients seen at JHH in the Center for Peripartum Optimization (CPO) clinic between January 2017 to January 2018 and comparing outcome data with a matched controlled group patients not seen at the CPO clinic. This matched controlled parturient group will be identified utilizing the JHH EMR and ICD-10 comorbidity codes.
  These patients will be female of child-bearing age that fits into the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | 1 year
  Total days of hospital admission

SECONDARY OUTCOMES:
Number of admissions from outside hospitals | 1 year
  The total number of admissions to any other hospitals prior to admission or after discharge
ICU admissions | 1 year
  Whether patient needed ICU admission or transfer
Opioids use | 1 year
  To determine if patient require opioid use
Neonatal Intensive Care Unit (NICU) admissions | 1 year
  Number of times a neonate got admitted to the NICU
Patient satisfaction | 1 year
  Whether patient was satisfied (yes/no) with treatment course based on survey filled out by patient.
Cost of inpatient admission | 1 year
  the entire admission cost of admission during hospital stay
Cost of outpatient care | 1 year
  The cost for outpatient care incurred by patient
Hospital readmissions rate | 1 year
  The number of times a patient got readmitted after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jamie D Murphy, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No